CLINICAL TRIAL: NCT00489606
Title: Clinical Trial to Investigate the Influence of Drug Interaction After Oral Administration of Tamsulosin and SK3530 in Healthy Male Volunteers
Brief Title: Phase I Study to Investigate the Drug Interaction After Oral Administration of Tamsulosin and SK3530
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SK3530_DI_TS
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Erectile Dysfunction
Keywords: SK3530; tamsulosin; hemodynamic interaction; safety
MeSH Terms: conditions — Erectile Dysfunction | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SK3530

SUMMARY:
To assess the pharamcodynamic effects of coadministrated SK3530(PDE5 inhibitor) and tamsulosin, phase I study in healthy volunteers was designed.

DETAILED DESCRIPTION:
During each of the two periods of a randomized, double-blind, placebo-controlled, crossover study, 16 healthy men received tamsulosin 0.2 mg daily for 7 days and either a single 100 mg of SK3530 or placebo on day7. The blood pressure and heart rate were monitored before and for 24 hours after SK3530 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* ages 20 to 50
* body weight of IBM±20%

Exclusion Criteria:

* cardiovascular disease
* color-blindness or weakness
* hypotension, hypertension, orthostatic hypertension
* abmormal QTc (>430 ms)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Maximal decrease from baseline in supine SBP | within 6 hrs after SK3530 or placebo

SECONDARY OUTCOMES:
Maximal decrease from baseline in standing SBP, supine/standing DBP & HR | within 6 hrs after SK3530 or placebo
Outlier analysis: i) Standing/supine SBP < 85 mmHg, DBP < 45 mmHg; ii) Change in standing/supine SBP > 30 mmHg, DBP > 20 mmHg | within 6 hrs after SK3530 or placebo
Incidence of postural hypotension | within 6 hrs after SK3530 or placebo

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Chang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea